CLINICAL TRIAL: NCT07252167
Title: A Comparative Evaluation of Clinical Outcomes and Cone-Beam Computed Tomography Findings of Enamel Matrix Derivative and Amniotic Membrane in Regenerative Endodontic Treatment of Non Vital Immature Permanent Anterior Teeth: A Randomized Clinical Trial
Brief Title: Comparison Between Emdogain and Amniotic Membrane as a Scaffold in Endodontic Regeneration of Immature Anterior Teeth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abrar Hamed Habib Yousef, Assistant Lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endodontic regeneration
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Non-vital Immature Anterior Teeth
Keywords: Revascularization, endodontic regeneration, Immature
MeSH Terms: interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Regenerative endodontic treatment using MTA (Experimental): Regenerative endodontic treatment with conventional blood clot technique.
  Interventions: Other: Regenerative endodontic treatment with conventional blood clot technique.
- Regenerative endodontic treatment using emdogain (Experimental): regenerative endodontic treatment with emdogain
  Interventions: Other: regenerative endodontic treatment with emdogain.
- Regenerative endodontic treatment using amniotic membrane (Other): regenerative endodontic treatment with amniotic membrane
  Interventions: Other: regenerative endodontic treatment with amniotic membrane

INTERVENTIONS:
Other: Regenerative endodontic treatment with conventional blood clot technique. — After local anesthesia, rubber dam isolation and access cavity preparation, pulp tissue extirpation/debridement, the root canal system is minimally instrumented. Copious irrigation is performed, gently with single-side vented needles. Canals are dried with paper points. Metapaste is injected as intracanal medication. At second session, check for absence of signs/symptoms. Copious gentle irrigation and drying of canals with paper points is done. Bleeding is created in root canal by over-instrumentation until bleeding is evident in the cervical portion of the canal. A lightly moistened sterile cotton pellet is placed into the canal, 3-4 mm apical to the CEJ, for 7-10 minutes to allow blood clot formation. Placement of MTA over the blood clot as a capping material. A 3-4 mm layer of glass ionomer is gently placed over the capping material. Followed by resin composite restoration.
  Arms: Regenerative endodontic treatment using MTA
Other: regenerative endodontic treatment with emdogain. — • After local anesthesia, rubber dam isolation and access cavity preparation, pulp tissue extirpation/debridement, the root canal system is minimally instrumented. Copious irrigation is performed, gently with single-side vented needles. Canals are dried with paper points. Metapaste is injected as intracanal medication. At second session, check for absence of signs/symptoms. Copious gentle irrigation and drying of canals with paper points is done. Bleeding is created in root canal by over-instrumentation until bleeding is evident in the cervical portion of the canal. A lightly moistened sterile cotton pellet is placed into the canal, 3-4 mm apical to the CEJ, for 7-10 minutes to allow blood clot formation. Emdogain is injected inside the canal on the blood clot up to the CEJ to act as a matrix for the cells. Placement of MTA over the blood clot as a capping material. A 3-4 mm layer of glass ionomer is gently placed over the capping material. Followed by resin composite restoration.
  Arms: Regenerative endodontic treatment using emdogain
Other: regenerative endodontic treatment with amniotic membrane — - After local anesthesia, rubber dam isolation and access cavity preparation, pulp tissue extirpation/debridement, the root canal system is minimally instrumented. Copious irrigation is performed, gently with single-side vented needles. Canals are dried with paper points. Metapaste is injected as intracanal medication. At second session, check for absence of signs/symptoms. Copious gentle irrigation and drying of canals with paper points is done. Bleeding is created in root canal by over-instrumentation until bleeding is evident in the cervical portion of the canal. A lightly moistened sterile cotton pellet is placed into the canal, 3-4 mm apical to the CEJ, for 7-10 minutes to allow blood clot formation. Amniotic membrane will adapted inside the canal on the blood clot up to the CEJ. Placement of MTA over the blood clot as a capping material. A 3-4 mm layer of glass ionomer is gently placed over the capping material. Followed by resin composite restoration.
  Arms: Regenerative endodontic treatment using amniotic membrane

SUMMARY:
To evaluate the clinical outcomes and cone-beam computed tomography findings of enamel matrix derivative and amniotic membrane in regenerative endodontic treatment of non-vital immature permanent anterior teeth

DETAILED DESCRIPTION:
To evaluate the clinical outcomes and cone-beam computed tomography findings of enamel matrix derivative in comparison to amniotic membrane and MTA as a conventional group in regenerative endodontic treatment of non-vital immature permanent anterior teeth

ELIGIBILITY:
Inclusion Criteria:

•Patients age ranges between 7 and 12 years at the time of enrolment including both genders. •Provision of informed consent by one parent or legal guardian. •At least one immature permanent anterior tooth diagnosed with pulp necrosis with or without periapical lesions. •Restorable teeth. •Compliant patient/parent. •Radiologic evidence of open apices (Teeth are considered immature when a minimum of 1 mm apical foramen width is evident)

Exclusion Criteria:

•Teeth with root fractures or split roots. •Presence of root resorptions. •Presence of periodontal pockets. •Developmental anomalies. •Presence of periapical radiolucency of more than 10 mm. •Tooth with class III mobility.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment of root length by CBCT | Baseline (immediately post-operative), an 12 months post-operative.
  For all cases, CBCT was taken at a setting of 3-7 mA and 120 kVp and an exposure time of 9 s. Each scan was taken over 360º with a 0.3 mm voxel size. The root length was measured using the CBCT ruler to draw a line from the center point of the line connecting CEJ to the most apical point in the center of the root apex (proximally and facially). The percentage of increase in root length was calculated using this formula:
  (12 months value - preoperative value )/Preoperative value X 100%
Radiographic assessment of diameter of apical foramen by CBCT | Baseline(immediately post-operative), and 12 months post-operative.
  Diameter of the apical foramen was measured using the CBCT ruler at the most apical points buccolingually at the sagittal (proximal) view of CBCT. It was also measured at the most apical points mesiodistally at the coronal (facial) view of CBCT. The percentage reduction of the apical diameter was calculated using this formula:
  ( preoperative value - 12-month value ) /Preoperative value *100%
Radiographic assessment of root area by CBCT | Baseline (immediately post-operative), and 12 months post-operative.
  Radiographic root area (RRA) was measured using a method described by Flake et al using the polygon selection tool of CBCT. Below a straight line marking the CEJ, the root area was outlined from the surrounding periodontal environment. Then, the pulp space area was measured by the same method using the polygon tool by tracing the reference points surrounding the pulp space. Finally, RRA was calculated by subtraction of the pulp space area from the outer root area. These measurements were made at proximal and facial views of CBCT . The percentage increase in RRA was calculated using this formula:
  ( 12-month value - preoperative value )/Preoperative value X 100 %
Radiographic assessment of size of periapical lesion by CBCT | Baseline (Immediately post-operative), and 12 months post-operative.
  Lesion size was measured by tracing the periphery of the lesion using the polygon tool of the CBCT from proximal and facial views of the CBCT. A closed polygon tool was used to delimit the border of the lesion to measure the area of the periapical lesion in (mm2).The percentage reduction of lesion size was calculated as follows:
  ( preoperative value - 12-month value ) /Preoperative value X 100 %

SECONDARY OUTCOMES:
Clinical assessment of presence/ absence of pain | Baseline, 3 months, 6 months, and 12 months post operative.
  Assessment of symptoms of patient whether there is a pain or not in each follow up period.
Clinical assessment of presence/ absence of mobility of teeth | Baseline, 3 months, 6 months, and 12 months post operative.
  Assessment of teeth whether they exhibit mobility or not
Clinical assessment of presence/ absence of associated sinus tract or swelling. | Baseline, 3 months, 6 months, and 12 months post operative.
  Assessment of teeth whether they exhibit associated sinus tract or swelling or not
Clinical assessment of presence/ absence of tenderness to palpation of adjacent soft tissues. | Baseline, 3 months, 6 months, and 12 months post operative.
  Assessment of teeth whether they exhibit tenderness to palpation of adjacent soft tissues or not
Clinical assessment of presence/ absence of tenderness to percussion | Baseline, 3 months, 6 months, and 12 months post operative.
  Assessment of teeth whether they exhibit tenderness to percussion

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes